CLINICAL TRIAL: NCT07073027
Title: Evaluating the Impact of Digital Media on Patient-Reported Experience and Outcomes in Pediatrics
Brief Title: How Digital Media Affects Kids' Healthcare Experiences and Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, John Jacob, Adjunct Professor, British Columbia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H24-00446
Record Dates: First submitted 2025-06-24; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Children; Adolescent; Anxiety; Pain; Education; Exposure; Virtual Reality
Keywords: pre-procedural anxiety; exposure therapy; virtual reality; education; children and adolescents; gamification
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2D video on phone (Active Comparator): In the 2D video arm, participants will see still images of the procedural room and tools / medical equipment that are played in a video. Each video contains a series of still images of the procedure room and stills of tools / medical equipment used in the procedure room (e.g., cast saw for the cast removal procedure, a coil for the MRI scan, etc.). As the narrator describes each tool / medical equipment an enlarged image of that tool medical equipment appears along with text. The participants randomized into this arm will hear the same audio as the other 2 arms (360 video, 360 video in VR). The difference in this group is that participants cannot interact with their media (i.e., they cannot swipe their smart phone or move their phone to look around the procedural room unlike the 360 video groups).
  Interventions: Other: 2D video on smartphone
- 360 video on phone without virtual reality (Active Comparator): In the 360 video arm, participants will see a still image of the procedural room played in a video format. Each video contains a single still 360 image of the procedure room and the tools / medical equipment used in the procedure room (e.g., cast saw for the cast removal procedure, a coil for the MRI scan, etc.). As the narrator describes each tool / medical equipment an enlarged image of that tool medical equipment appears at the side of the tool / medical equipment along with text (similar to the 2D video). The participants randomized into this arm will hear the same audio as the other 2 arms (2D video, 360 video in VR). The difference in this group is that participants can interact with their media (i.e., they can swipe their smart phone using their finger to see an entire 360 view of the procedural room, but unlike the 360 VR group, this 360 group will not be using it the VR headset).
  Interventions: Other: 360 video on smartphone inserted into VR cardboard headset
- 360 video on phone in virtual reality (Experimental): In the 360 video in virtual reality arm, participants will see a still image of the procedural room played in a video format. Each video contains a single still 360 image of the procedure room and the tools / medical equipment used in the procedure room (e.g., cast saw for the cast removal procedure, a coil for the MRI scan, etc.). As the narrator describes each tool / medical equipment an enlarged image of that tool medical equipment appears at the side of the tool / medical equipment along with text (similar to the 2D video). The participants randomized into this arm will hear the same audio as the other 2 arms (2D video, 360 video in VR). The difference in this group is that participants can interact with their media using a VR headset (i.e., they can move their head, or physically turn around which moves the point of view of the video and thus their view of the procedural room).
  Interventions: Other: 360 video on smartphone

INTERVENTIONS:
Other: 2D video on smartphone — 2D video with audio viewed on smartphone
  Arms: 2D video on phone
Other: 360 video on smartphone — 360 video with audio viewed on smartphone (not in virtual reality)
  Arms: 360 video on phone in virtual reality
Other: 360 video on smartphone inserted into VR cardboard headset — 360 video with audio in virtual reality
  Arms: 360 video on phone without virtual reality

SUMMARY:
The goal of this clinical trial is to learn whether different forms of media (2D, 360, or 360 in virtual reality) have different impacts on pre-procedural anxiety and post-procedural pain in children. The main questions it aims to answer are:

Does one type (and richness) of media reduce pre-procedural anxiety and post-procedural pain more than another type of media? For example, will learning about an upcoming procedure by watching a 360 video in virtual reality reduce pre-procedural anxiety more than learning about the same upcoming procedure by watching it in a 2D video or 360 video?

The second question is whether watching a 360 video in VR about an upcoming procedure more effective in reducing pre-procedural anxiety and post-procedural pain compared to the 2D video or the 360 video without VR groups for specific procedures? For example, is watching an explanation of a procedure in VR always more effective in reducing pre-procedural anxiety and post-procedural pain, or is it procedure specific (i.e., watching a video about surgery preparation is more effective in VR, but for cast removal it doesn't matter whether participants learn about their procedure viewed through VR, 360 video, or 2D)?

DETAILED DESCRIPTION:
Children experience anxiety before medical procedures, which have negative effects. Educating them about what to expect can help reduce this anxiety. In this study, the investigators aim to prepare children for procedures using 2D and 360 video with audio, including virtual reality (VR). Children and adolescents aged 5-18 and adults aged 19-23 will be randomized to receive either 2D video with audio-, 360 video with audio-, or 360 video with audio in VR-based preparation materials. Participants will complete patient-reported outcomes and experience surveys before and after their preparation through a secure mobile app, accessible through their smartphone. The investigators hypothesize that VR video-based education will reduce anxiety and improve patient experience compared to when patients learn about their procedure through a 2D video with audio and a 360 video with audio without VR. The investigators further hypothesize that the media fidelity, in terms of level of immersiveness, will have an effect on associated outcomes.

In this study the investigators plan to recruit 500 participants between the ages of 5 to 23. Participants will be randomized into one of 3 preparation groups (e.g., 2D video w/ audio, 360 video w/ audio w/o VR, or 360 video w/ in VR). Participants in the 2D video-preparation group will watch and hear descriptions about the hospital environment, equipment, staff, and / or their scheduled upcoming procedure. Participants in the 360 video with audio-based preparation group will also see and hear descriptions of the hospital environment, equipment, staff, and / or their scheduled upcoming procedure. However, unlike the 2D video-based group, 360 video group will have the ability to swipe on their phone and see 360 views of the environment (i.e., the procedure room). Participants in the 360 video with audio in VR-based preparation group will see and hear videos of the hospital environment, equipment, staff, and /or their scheduled upcoming procedure in VR. Participants randomly assigned to this group will have the ability to move their head around using a cardboard VR headset and see 360 views of the hospital environment. Each participant will have their media tailored to their specific procedure. For example, participants that are undergoing a cast removal will be given different media (i.e., cast removal specific material) compared to someone who is scheduled to receive a magnetic resonance imaging scan. Participants will use their preparation materials at least once, approximately 1 week prior to their scheduled procedure.

Participants (i.e., patients) will take a series of short surveys before and after experiencing their preparation material. Surveys will include self-report anxiety and pain measures. After the procedure, the investigators plan to follow-up with the participants at 3 separate occasions. During follow-up assessments the investigators will ask participants about their anxiety as well as pain. The patient's caregivers will also complete baseline state and trait anxiety measures in addition to a satisfaction survey, but all other surveys / measures will be completed by the patient (i.e., child).

Interested participants will first complete an online screening survey to ensure their eligibility on Qualtrics. Upon successful screening, the user will be allowed to proceed to the consent and assent agreement page on Qualtrics. After consent and assent, participants will complete baseline survey data (demographics, trait anxiety) on Qualtrics. After baseline survey data, the study team will email the user to a link to where participants will be asked to download and register (password, and e-mail address) to access the app. In this way, data collected in the app will be de-identified but linked to the consent form data that is collected on Qualtrics via a randomly generated number that will be recorded by the app. All intervention media (2D video with audio, 360 video with audio w/o VR, and 360 video with audio in VR) will be accessed through the secure app (in compliance with local and provincial/national data collection/residency policies). This app will need to be downloaded. Upon successful registration, the research team will provide them with a unique code. The code will allow participants to enter into the app and the appropriate room where their material is located. Because Qualtrics is embedded within the app, participants will complete surveys within the app but through Qualtrics.

To access the media (2D video with audio, 360 video with audio on smartphone, or 360 video with audio viewed in VR) participants will explore a gamified version of the BC Children's Hospital. Participants will create an avatar and set a procedure date before leaving the home room (i.e., a bedroom). After setting a procedure date, participants will be able to access the lobby of the hospital and their procedure room (provided that it is within 7 days of their scheduled procedure). The gamified hospital environment is modeled after BC Children's Hospital and included non-playable characters, a learning kiosk, and a computer to finish surveys.

For those randomized to receive the 360 video-based preparation, participants will receive standard-of-care specific to the division/clinic that scheduled their procedure, with audio-based descriptions of their upcoming procedure, as well as videos. Videos will contain a voice-over tour and procedural experience, specific to the participant's procedure, including an orientation to the hospital environment, equipment, and sometimes each procedural step specific to their procedure. Thus, there will be multiple 360 video-based exposure and education videos, each one specific to the procedure the participant is scheduled to have. Participants randomized to the 360 video with audio WITHOUT VR, will watch the videos on their phone without the use of a VR headset. They will be able to swipe on their phone and move the video around to fully experience the hospital environment. Participants randomized to the immersive arm of the study (e.g., VR), will be able to view video in virtual reality with the use of a VR-viewer / headset that utilizes their existing mobile phone. The VR headset will be provided to participants at the time of recruitment or sent to them through mail.

Participants in the 2D video with audio-based group will receive standard-of-care specific to the division/clinic that scheduled their procedure plus 2D video with audio-based preparation. 2D video with audio-based preparation will include and spoken descriptions of the hospital environment, the staff, equipment, and / or each procedural step specific to their procedure. Therefore, persons that are in the 2D video with audio-based preparation group will receive the same information as the 360 video groups, however, all exposure / education will be in a 2D video format (image stills played in a video) that is specific to the procedure the participant is scheduled to have. Therefore, there will be multiple 2D video with audio-based exposure scenarios, each one specific to the procedure the participant is scheduled to have.

All participants will use a standalone mobile app to access their preparation media. It should be noted that all participants will have the opportunity to access a VR tutorial as a part of their participation in this study. Participants that are not randomized to the immersive video arm will not be able to access content specific to their procedure, but instead will be able to experience a VR environment briefly within the gamified version of the hospital. All participants will be able to do this.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5 to 23
* Able to follow instructions and communicate in English
* Own or have access to a smartphone
* Scheduled for an upcoming (approved) procedure.

Exclusion Criteria:

* Under the age of 5 or older than 23
* Vision, hearing, cognitive, and/or motor impairments
* Cannot follow instructions and/or communicate in English
* Do not own or have access to a smartphone.

Ages: 5 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline (immediately before the intervention)
  Measurement of anxiety. To measure state anxiety we are using the number 0-10 anxiety score. The scale goes from 0 to 10 with 10 being the worst imaginable anxiety.
Anxiety | Periprocedural (immediately after the intervention)
  Measurement of anxiety. To measure state anxiety we are using the number 0-10 anxiety score. The scale goes from 0 to 10 with 10 being the worst imaginable anxiety.
Anxiety | 1 day after procedure
  Measurement of anxiety. To measure state anxiety we are using the number 0-10 anxiety score. The scale goes from 0 to 10 with 10 being the worst imaginable anxiety.
Anxiety | 1 week after procedure
  Measurement of anxiety. To measure state anxiety we are using the number 0-10 anxiety score. The scale goes from 0 to 10 with 10 being the worst imaginable anxiety.
Anxiety | 4 weeks after procedure
  Measurement of anxiety. To measure state anxiety we are using the number 0-10 anxiety score. The scale goes from 0 to 10 with 10 being the worst imaginable anxiety.

SECONDARY OUTCOMES:
Pain intensity | Baseline (immediately before the intervention)
  Measurement of pain using numeric rating scale of pain. The scale goes from 0 to 10 with 10 being the worst hurt you could possibly imagine.
Pain intensity | Periprocedural
  Measurement of pain using numeric rating scale of pain. The scale goes from 0 to 10 with 10 being the worst hurt you could possibly imagine.
Pain intensity | 1 day after procedure
  Measurement of pain using numeric rating scale of pain. The scale goes from 0 to 10 with 10 being the worst hurt you could possibly imagine.
Pain intensity | 1 week after procedure
  Measurement of pain using numeric rating scale of pain. The scale goes from 0 to 10 with 10 being the worst hurt you could possibly imagine.
Pain intensity | 4 weeks after the procedure
  Measurement of pain using numeric rating scale of pain. The scale goes from 0 to 10 with 10 being the worst hurt you could possibly imagine.

OTHER OUTCOMES:
Ready for procedure and recommendation | Periprocedural (immediately after the intervention)
  In the post-intervention survey, we ask both the patients and caregivers whether they think they and their child is ready for the upcoming procedure, respectively. We ask the patient "Do you feel ready for your [procedure]?" with the option of "No", "Maybe", and "Yes". We also ask the patient "Pretend a family member or friend is going to have surgery like you. How likely are you to tell your family or friends about this app?" on a 0 to 10 scale with 0 labeled as "Not at all likely" and a 10 labeled as "Extremely likely". We also ask the parent / guardian, "To what extent do you think your child is ready for their procedure?" with the option of "Not at all prepared", "Somewhat prepared", "Fully prepared". We also ask the parent / guardian "How likely are you to recommend the app to other families or friends with children undergoing the same procedure?" on a 0 to 10 scale with 0 labeled as "Not at all likely" and 10 labeled as "Extremely likely".
Procedure satisfaction and recommendation follow-up | 1 day after procedure
  We ask both the patients and parent about the procedure. We ask the patient "How did the procedure go?" with the option of "Very good", "Good", "Bad" and "Very bad". We also ask the patient and the parent "Were your prepared for your procedure?" with the option of "Yes", "No", and "I don't know". We also ask "Pretend a family member or friend is going to have surgery like you. How likely are you to tell your family or friends about this app?" on a 0 to 10 scale with 0 labeled as "Not at all likely" and a 10 labeled as "Extremely likely". We also ask the parent, "Overall, how satisfied are you with how the procedure went?" with the option of "Very dissatisfied", "dissatisfied", "Neutral ", "Satisfied", "Very Satisfied" and "N/A". We also ask the parent "How likely are you to recommend the app to other families or friends with children undergoing the same procedure?" on a 0 to 10 scale with 0 labeled as "Not at all likely" and 10 labeled as "Extremely likely".

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT07073027/Prot_SAP_000.pdf